CLINICAL TRIAL: NCT04259229
Title: Mediterranean Diet and Mushrooms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Mushroom Council (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Principal Investigator, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IRB-2019-650
Record Dates: First submitted 2019-12-19; First posted 2020-02-06 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Diet, Healthy
Keywords: Mediterranean; Mushrooms

STUDY DESIGN:
Intervention Model Description: For this investigator-blinded, randomized, parallel design study, 100 participants (60 to finish; n=30/group) will complete a 10-week study period, which includes a 2-week baseline testing period (no diet control), followed by an 8-week controlled diet period (Figure 1). In order to define the effects of adding mushrooms to a healthy dietary pattern on fasting blood glucose and insulin concentrations and blood pressures, we will provide a Mediterranean-style diet devoid of mushrooms as the control diet for this study. Questionnaires assessing depression/anxiety, perceived quality of life, and mood will be administered and the results will provide a foundation to power future, more robust, studies.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mushroom intervention (Experimental): Subjects will be randomized and assigned to consume the Mediterranean Diet with mushrooms for eight weeks.
  Interventions: Other: Mediterranean Diet -- Mushrooms
- Control (Active Comparator): Subjects will be randomized and assigned to consume the Mediterranean Diet without mushrooms for eight weeks.
  Interventions: Other: Mediterranean Diet -- Control

INTERVENTIONS:
Other: Mediterranean Diet -- Mushrooms — During the 2-week baseline period all participants will consume their usual, unrestricted self-chosen diets. During intervention weeks 1-8, all participants will consume the same Mediterranean-style diet, rich in fruits and seafoods and lower in dairy, designed to meet their estimated energy needs. The mushroom group will consume 0.5 cups/day of cooked mushrooms (white button mushrooms and yellow oyster mushrooms on 4 and 3 days/week, respectively). All foods will be provided to subjects during the intervention to achieve the desired eating pattern.
  Arms: Mushroom intervention
Other: Mediterranean Diet -- Control — During the 2-week baseline period all participants will consume their usual, unrestricted self-chosen diets. During intervention weeks 1-8, all participants will consume the same Mediterranean-style diet, rich in fruits and seafoods and lower in dairy, designed to meet their estimated energy needs. The control group will not consume mushrooms at any point. All foods will be provided to subjects during the intervention to achieve the desired eating pattern.
  Arms: Control

SUMMARY:
The investigators propose to assess the effects of including mushrooms as part of a healthy eating pattern on indices of perceived mental health/anxiety/depression, along with risk factors for cardiovascular disease and type 2 diabetes.

DETAILED DESCRIPTION:
The investigators hypothesize that consuming mushrooms as part of a healthy eating pattern will lead to greater improvements in fasting insulin concentrations and systolic and diastolic blood pressures. The brain health-related outcomes and other cardiometabolic risk outcomes (e.g. lipoprotein particle size) are exploratory due to the paucity of human research addressing these important topics. Collectively, this short-term (8-week) randomized, controlled feeding trial will provide important pilot data to inform the plausibility, focus, and design of longer-term intervention trials, consistent with The Mushroom Council's research agenda.

ELIGIBILITY:
Inclusion Criteria:

* Male or female;
* age 30-69 y;
* BMI: 25.0-34.9 kg/m2;
* Not severely or extremely depressed (Beck's Depression Inventory score ≤30)
* Total cholesterol <240 mg/dL, low-density lipoprotein cholesterol <160 mg/dL, triglycerides <400 mg/dL, fasting glucose <110 mg/dL;
* Systolic/diastolic blood pressure <140/90 mm Hg;
* Body weight stable for 3 months prior (± 3 kg);
* Stable physical activity regimen 3 months prior;
* Medication use stable for 6 months prior;
* Non-smoking;
* Non-diabetic;
* Not acutely ill;
* Females not pregnant or lactating;
* Participants must be willing and able to consume the prescribed diets and travel to testing facilities.

Exclusion Criteria:

* BMI <25 or >35;
* Severely depressed (Beck's Depression Inventory score >30);
* Total cholesterol >240 mg/dL, low-density lipoprotein cholesterol >160 mg/dL, triglycerides >400 mg/dL, fasting glucose >110 mg/dL;
* Body weight changes in previous 3 months (±3 kg);
* Changes in physical activity regimen in the previous 3 months;
* Medication changes in the previous 6 months;
* Smoking;
* Diabetic;
* Acute illness;
* Pregnant or lactating;
* Allergic to mushrooms

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Change in perceived depression from baseline to post-intervention | 8 weeks
  Beck's Depression Inventory questionnaire
Change in perceived depression from baseline to post-intervention | 8 weeks
  Patient Health Questionnaire-9
Change in perceived anxiety from baseline to post-intervention | 8 weeks
  General Anxiety Disorder-7 questionnaire
Change in cognitive function from baseline to post-intervention | 8 weeks
  Repeatable Battery for the Assessment of Neuropsychological Status
Change in perceived daily mood from baseline to post-intervention | 8 weeks
  Profile of Mood States
Change in perceived quality of life from baseline to post-intervention | 8 weeks
  Medical Outcomes Study 36-Item Short Form Health Survey Version 2
Risk factors for cardiovascular disease | 8 weeks
  Blood pressure
Risk factors for cardiovascular disease | 8 weeks
  Complete metabolic panel
Risk factors for cardiovascular disease | 8 weeks
  Lipoprotein Particle Plus (LPP+) Panel
Risk factors for type 2 diabetes | 8 weeks
  Complete metabolic panel
Change in immunity/inflammation markers | 8 weeks
  Complete Cytokine 13 Panel -- all outcomes reported as pg/mL
Change in immunity/inflammation markers | 8 weeks
  Complete Immunoglobulin Panel -- all outcomes reported as mg/dL

SECONDARY OUTCOMES:
Body weight | 8 weeks
  Measures of weight (kg)
Gut microbiota | 8 weeks
  Stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Wayyne Campbell, PhD, Principal Investigator — Purdue University
Locations (2):
- United States (2):
  - Purdue University, West Lafayette, Indiana
  - Purdue University - Stone Hall 700 W State St, West Lafayette, Indiana

REFERENCES:
- [Derived] Uffelman CN, Schmok JN, Campbell RE, Hartman AS, Olson MR, Anderson NL, Reisdorph NA, Tang M, Krebs NF, Campbell WW. Consuming Mushrooms When Adopting a Healthy Mediterranean-Style Dietary Pattern Does Not Influence Short-Term Changes of Most Cardiometabolic Disease Risk Factors in Healthy Middle-Aged and Older Adults. J Nutr. 2024 Feb;154(2):574-582. doi: 10.1016/j.tjnut.2023.12.026. Epub 2023 Dec 20. PMID 38135005